CLINICAL TRIAL: NCT01667289
Title: A Randomized Phase II Study of Comparing Radiotherapy Alone With Concurrent Chemoradiation in Patients With Low Risk NK/T-cell Lymphoma
Brief Title: Radiotherapy Alone Versus Concurrent Chemoradiation in Low Risk NK/T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpected high grade of mucositis observed
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Assocaite Director of Medical Oncology Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 12-01
Record Dates: First submitted 2012-08-13; First posted 2012-08-17 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: NK/T-cell lymphoma; Methotrexate; Radiotherapy; Concurrent chemoradiation
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy alone (Active Comparator): Radiotherapy alone Technique: IMRT Total Dose: 50 Gy Per fraction: 2 Gy
  Interventions: Radiation: Radiotherapy alone
- Concurrent chemoradiation (Experimental): Concurrent chemoradiation
  Chemotherapy:
  Methotrexate 40 mg/m2 weekly X 5 Radiotherapy Technique: IMRT Total dose: 50 Gy Per Fraction: 2 Gy
  Interventions: Radiation: Radiotherapy alone; Drug: Concurrent chemoradiation

INTERVENTIONS:
Radiation: Radiotherapy alone — Radiotherapy alone Technique: IMRT Total Dose: 50 Gy Per fraction: 2 Gy
Drug: Concurrent chemoradiation — Concurrent chemoradiation
  Chemotherapy:
  Methotrexate 40 mg/m2 weekly X 5 Radiotherapy Technique: IMRT Total dose: 50 Gy Per Fraction: 2 Gy
  Other Names: MTX
  Arms: Concurrent chemoradiation

SUMMARY:
The purpose of this study is to prove the superiority of concurrent chemoradiation compared with radiotherapy alone in patients with low risk NK/T-cell lymphoma.

DETAILED DESCRIPTION:
Radiotherapy alone is commonly used in NK/T-cell lymphoma without adverse risk including lymph node involvement, local invasion, B symptoms and high LDH level. Recently, methotrexate was prove to be a radiosensitizer in NK/T-cell lymphoma cells. Therefore, the investigators aim to verify the superiority and safety of weekly methotrexate in combination with radiotherapy in a randomized phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-75 years old
* Histological confirmed, previously untreated stage IE nasal NK/T cell lymphoma without following risk factors including local invasion, B symptoms and high LDH level
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Adequate bone marrow and organ functions

Exclusion Criteria:

* non-nasal NK/T-cell lymphoma
* Prior exposure of methotrexate
* With third space effusion
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
3-year Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall response rate | 3 years
3-year overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China